CLINICAL TRIAL: NCT01339312
Title: Immunogenicity and Safety of the Purified Vero Rabies Vaccine - Serum Free in Comparison With the Reference Purified Vero Rabies Vaccine in Post-exposure Use in Healthy Subjects in China
Brief Title: Study of the Purified Vero Rabies Vaccine - Serum Free in Comparison With the Reference Purified Vero Rabies Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VRV08; U1111-1117-7193 (Other: WHO)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Rabies; Rabies Virus
Keywords: Rabies; Rabies virus; Purified Vero Rabies Vaccine - Serum Free
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VRVg Vaccine Group 1 (Experimental): Participants aged 18 years or older will receive Purified Vero Rabies Vaccine Serum Free (VRVg)
  Interventions: Biological: Purified inactivated rabies vaccine, serum free
- VRVg Vaccine Group 2 (Experimental): Participants aged 10 to 17 years will receive Purified Vero Rabies Vaccine Serum Free (VRVg)
  Interventions: Biological: Purified inactivated rabies vaccine, serum free
- Verorab Vaccine Group 1 (Active Comparator): Participants aged 18 years or older will receive Verorab Vaccine
  Interventions: Biological: Purified Vero Rabies Vaccine
- Verorab Vaccine Group 2 (Active Comparator): Participants aged 10 to 17 years will receive Verorab Vaccine
  Interventions: Biological: Purified Vero Rabies Vaccine

INTERVENTIONS:
Biological: Purified inactivated rabies vaccine, serum free — 0.5 mL, Intramuscular
  Other Names: Purified Vero Rabies Vaccine Serum Free
  Arms: VRVg Vaccine Group 1
Biological: Purified inactivated rabies vaccine, serum free — 0.5 mL, Intramuscular
  Other Names: Purified Vero Rabies Vaccine Serum Free
  Arms: VRVg Vaccine Group 2
Biological: Purified Vero Rabies Vaccine — 0.5 mL, Intramuscular
  Other Names: Verorab Vaccine
  Arms: Verorab Vaccine Group 1
Biological: Purified Vero Rabies Vaccine — 0.5 mL, Intramuscular
  Other Names: Verorab Vaccine
  Arms: Verorab Vaccine Group 2

SUMMARY:
This study is designed to gather safety and immunogenicity data with Purified Vero Rabies Vaccine - Serum Free (VRVg), when given in a post-exposure prophylaxis vaccination schedule, using the Essen regimen, across different populations.

Primary Objective:

* To demonstrate that VRVg is at least as immunogenic as the reference vaccine, Verorab vaccine, in terms of proportion of participants with a rabies virus neutralizing antibody titer ≥ 0.5 IU/mL at Day 14, i.e., before the fourth vaccination, in participants aged 10 to 17 years and in participants aged 18 years and over.

Secondary Objectives:

* To assess the clinical safety of VRVg after each vaccination when administered in a post-exposure prophylaxis vaccination schedule in each respective age group and overall
* To describe the immune response induced by VRVg before the fourth vaccination and 14 days after the last vaccination in each respective age groups and overall.

DETAILED DESCRIPTION:
All participants will receive five vaccinations (on Days 0, 3, 7, 14, and 28) and will be assessed for immunogenic response on Days 0, 14, and 42. They will also be monitored for safety from the day of the first vaccination and for up to 6 months after the final vaccination.

ELIGIBILITY:
Inclusion Criteria:

Adults (≥ 18 years)

* Aged ≥ 18 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination

Subjects aged 10-17 years:

* Aged 10 to 17 years on the day of inclusion
* Informed consent form has been signed and dated by the parent(s) or another legally acceptable representative and by subjects aged 12 years and over. In addition, provision of assent form signed by subjects aged 10 to 11 years
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures
* For a female of childbearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination, until at least 4 weeks after the last vaccination.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine during the course of the trial
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, or reported by the parent/guardian
* At high risk for rabies infection during the trial: (such as veterinarians and their staff, animal handlers, rabies researchers, and certain laboratory workers, persons whose activities bring them into frequent contact with rabies virus or potentially rabid bats, raccoons, skunks, cats, dogs, or other species at risk for having rabies, people travelling where rabies is enzootic, previous bite by a rabid animal with no post-exposure treatment administered)
* Known systemic hypersensitivity to any of the vaccine components , or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination, or reported by the parent/guardian
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator .

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Information on the rabies virus neutralizing antibody (RVNA) titer post vaccination | Day 14
  Rabies virus neutralizing antibody (RVNA) titer as determined by rapid fluorescent focus inhibition test (RFFIT)

SECONDARY OUTCOMES:
Information concerning the safety in terms of solicited injection site and systemic reactions, unsolicited adverse events, and serious adverse events post vaccination. | Day 1 up to 6 months post last vaccination
  Solicited Injection Site Reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Fever (Temperature), Headache, Malaise, Myalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Nanning, Guangxi, China

REFERENCES:
- [Result] Li R, Huang L, Li J, Mo Z, He B, Wang Y, Wu X, Minutello M, Guinet-Morlot F, Pichon S. A next-generation, serum-free, highly purified Vero cell rabies vaccine is safe and as immunogenic as the reference vaccine Verorab(R) when administered according to a post-exposure regimen in healthy children and adults in China. Vaccine. 2013 Dec 5;31(50):5940-7. doi: 10.1016/j.vaccine.2013.10.043. Epub 2013 Oct 19. PMID 24148575
- See also: Related Info — http://www.sanofipasteur.com